CLINICAL TRIAL: NCT05037461
Title: PRIME Study: Precision Radiotherapy Using MR-linac for Pancreatic Neuroendocrine Tumours in MEN1 Patients
Brief Title: Precision Radiotherapy Using MR-linac for Pancreatic Neuroendocrine Tumours in MEN1 Patients
Acronym: PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: J.M. de Laat (Other)
Collaborators: Radboud University Medical Center (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Leiden University Medical Center (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor-Investigator, J.M. de Laat, Principal Investigator (Md, PhD), UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77809.041.21
Record Dates: First submitted 2021-08-25; First posted 2021-09-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Neuroendocrine Tumor of Pancreas; Multiple Endocrine Neoplasia Type 1
MeSH Terms: conditions — Adenoma, Islet Cell; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-dose-high precision MR-guided radiotherapy (Experimental): Radiotherapy for pancreatic NET will be delivered in an image-guided, hypofractionated scheme of 5 fractions of 8 Gy, prescribed to 95% of the planning target volume (PTV). Treatment is delivered on alternate days 2 or 3 times a week with a maximum overall treatment time of 14 days on the 1.5T MR-Linac (Elekta Unity MR-Linac).
  The Gross Tumor Volume (GTV) is defines as the pNET visible on pre-treatment CT and MRI scan. No clinical target volume (CTV) is used. The PTV is made by adding a 3mm margin to the GTV.
  The treatment plan is a 9-14 field intensity modulated radiotherapy (IMRT) plan with dose prescribed to 95% of the PTV. While respecting the dose constraints to adjacent tissues
  Interventions: Radiation: High-dose-high precision MR-guided radiotherapy

INTERVENTIONS:
Radiation: High-dose-high precision MR-guided radiotherapy — MR-guided radiotherapy as described in the group information

SUMMARY:
Patients with the Multiple Endocrine Neoplasia type 1 (MEN1) syndrome are genetically predisposed for developping multiple pancreatic neuro-endocrine tumours (pNET). The management of small (pNET) in both MEN1 and sporadic cases, pose a major clinical challenge. At present, pancreatic surgery is the only curative treatment but it is associated with high morbidity. To reduce the morbidity ascosiated with surgery and thereby potentially improve quality of life for MEN1 patients introduction of less invasive techniques for treatment of pNET is important. High-dose-high precision MR-guided radiotherapy (MRgRT) holds promise as a new less invasive treatment option for pNET. The aim of this study is to assess efficiacy and safety of MRgRT for treatment of pNET in MEN1 patients.

DETAILED DESCRIPTION:
Background Patients with the Multiple Endocrine Neoplasia type 1 (MEN1) syndrome are genetically predisposed for developping multiple pancreatic neuro-endocrine tumours (pNET), with a cumulative pNET incidence of over 80% at an age of 80 years. In MEN1 patients, metastatic pNET is the primary cause of premature death.

The management of small (pNET) in both MEN1 and sporadic cases, pose a major clinical challenge. At present, pancreatic surgery is the only curative treatment. Since surgery is associated with significant short- and long-term morbidity the management of small pNET depends on carefully outweighing the risk of liver metastasis leading to premature death and the morbidity of pancreatic surgery. Guidelines advocate that for tumours smaller than 2 cm an intensive watchful waiting strategy seems to be safe. However, although most pNETs remain indolent for years, many lesions eventually progress and metastasize. To prevent the development of metastases for growing tumours or tumours above 2 cm a surgical resection is advised. Due to the high incidence of pNET in the MEN1 population many MEN1 patients receive surgery for pNET in their lifespan and cope with the morbidity of pancreatic surgery. To reduce the morbidity ascosiated with surgery and thereby potentially improve quality of life for MEN1 patients introduction of less invasive techniques for treatment of pNET is important.

High-dose-high precision MR-guided radiotherapy (MRgRT) holds promise as a new less invasive treatment option for pNET. With MRgRT accurate and precise delivery of high irradiation dose levels to the pNET is possible, while monitoring the tumor with MR imaging. The UMC Utrecht has pioneered the development of this technology, and gained experience with MRgRT treatments for patients with pancreatic adenocarcinoma and other upper abdominal malignancies.

Aim Aim of this project is to assess the safety and efficacy of high-dose-high precision MRgRT for pNET in a cohort of MEN1 patients that will require surgery in the near future.

Methods Efficacy and safety of MRgRT will be explored in a prospective cohort study of MEN1 patients with pNET, the Precision Radiotherapy using MRLInac for Pancreatic Neuroendocrine Tumours in MEN1 patients (PRIME)study. The PRIME study is a single arm interventional cohort study, recruiting 20 MEN1 patients enrolled in the Dutch MEN1 Study Groups (DMSG) longitudinal cohort. Eligible patients are patients with pNET surpassing 2.0 cm, and patients with a growing pNET measuring between 1.0- 2.0 cm. Patients who give informed consent will receive MRgRT with a minimum dose to the tumour bed of 40 Gy in 5 fractions delivered within 2 weeks. The primary outcome will be the change in maximum diameter of pNET at follow-up MRI scan at 12 months after diagnosis. Secondary outcome parameters include incidence of surgical resection following MRgRT, toxicity of radiotherapy, quality of life, endocrine and exocrine pancreatic functioning, metastases free survival, overall survival and tumour characteristics on follow-up MRI.

ELIGIBILITY:
All patients meeting the following criteria will be assessed for in the tumour board:

* lesions measuring between 2cm and 3cm.
* pNET lesions with a size between 1.0 and 2.0 cm and moderate growth of the lesion (2-4 mm/ year) on sequential follow-up scans.
* pNET lesions with a size between 1.0 and 2.0 cm and minimal growth of the lesion (1 mm/ year) reconfirmed on 3 or more sequential follow-up scans.
* Patients with in situ remaining 1.0 - 2.0 cm lesions after previous resection of a larger lesion.

All patients with such lesion and an indication for surgery are considered eligible for participation in the PRIME study.

Exclusion Criteria:

* Suspected malignant pNET as per the tumour board assessment, including the criteria:
* pNET lesions of more than 3 cm in size
* rapid growth of pNET lesions with more than 4mm per year
* Symptomatic pNET because of hormone production, with the exception of gastrinomas which are located in the submucosa of the duodenum
* concurrent treatment with a somatostatin analog
* concurrent treatment with chemotherapy
* peptide receptor radionuclide therapy in the past 12 months
* history of radiotherapy in the upper abdominal region
* MRI contraindications as per usual clinical care, such as claustrophobia and metal or electronic implants not compatible with MRI.
* Pregnancy
* (Other) metastatic disease
* WHO performance score 3-4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in tumor size | 12 months
  Change in maximal diameter of pNET measured at follow-up MRI

SECONDARY OUTCOMES:
Tumour progression | 12 months
  Number of patients with signs of growth or metastasis at follow-up
Pancreatic surgery | 12 months
  Number of patients that require surgical treatment following MRgRT
Toxicity of radiotherapy | 12 months
  Toxicity of radiotherapy graded according to Common Terminology Criteria for Adverse Events v4.0 scale
Health-related quality of life by SF-36 | 6 months, 12 months
  Short Form Health Survey 36 items
Health-related quality of life by Eq5D | 6 months, 12 months
  EuroQol 5D instrument
Health-related quality of life by PROMIS-29 | 6 months, 12 months
  PROMIS 29 profile
fasting glucose | 12 months
  fasting glucose in evaluation of endocrine and exocrine pancreatic function
blood cell count, | 12 months
  blood cell count in evaluation of endocrine and exocrine pancreatic function
serum iron | 12 month in evaluation of endocrine and exocrine pancreatic function
  serum iron v
vitamin B12 | 12 months
  vitamin B12 in evaluation of endocrine and exocrine pancreatic function
folate | 12 months
  folate in evaluation of endocrine and exocrine pancreatic function
faecal fat test | 12 months
  faecal fat test in evaluation of endocrine and exocrine pancreatic function
faecal trypsin | 12 months
  faecal trypsin in evaluation of endocrine and exocrine pancreatic function
faecal elastase | 12 months
  faecal elastase in evaluation of endocrine and exocrine pancreatic function
metastases free survival | 12 months
  Measured at follow-up imaging
overall survival | 12 months
  survival

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be placed in a repository and made available upon reasonable request, as stated in our data management plan.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon closure of the study database untill a minumum of 15 years
Access Criteria: Upon reasonable request